CLINICAL TRIAL: NCT02589522
Title: Phase 1 Trial to Determine the Recommended Phase 2 Dose (RP2D) of M6620 (VX-970, Berzosertib) When Combined With Whole Brain Radiotherapy (WBRT) in Patients With Brain Metastases From Lung Cancer
Brief Title: Testing the Safety of M6620 (VX-970) When Given With Standard Whole Brain Radiation Therapy for the Treatment of Brain Metastases From Non-small Cell Lung Cancer, Small Cell Lung Cancer, or Neuroendocrine Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01779; NCI-2015-01779 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HP-00068292; 9952 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 9952 (Other: CTEP); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186690 (NIH); UM1CA186691 (NIH)
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Lung Neuroendocrine Neoplasm; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Lung Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Brain; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Brain Neoplasms; Lung Neoplasms | interventions — berzosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (VX-970, whole-brain radiation therapy) (Experimental): Patients undergo whole-brain radiation therapy QD 5 days a week for 15 fractions. Patients also receive berzosertib IV over 60-90 minutes twice a week, 18-30 hours after first radiation therapy. Treatment continues for 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Berzosertib; Other: Quality-of-Life Assessment; Radiation: Whole-Brain Radiotherapy
- Group II (VX-970, surgery, whole-brain radiation therapy) (Experimental): Patients receive berzosertib IV over 60-90 minutes 2-4 hours prior to surgery. After surgery, patients undergo whole-brain radiation therapy and receive berzosertib as in Group I.
  Interventions: Drug: Berzosertib; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery; Radiation: Whole-Brain Radiotherapy

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Group II (VX-970, surgery, whole-brain radiation therapy)
Radiation: Whole-Brain Radiotherapy — Undergo whole-brain radiation therapy
  Other Names: WBRT; whole-brain radiation therapy

SUMMARY:
This phase I trial studies the side effects and best dose of berzosertib (M6620 [VX-970]) when given together with whole brain radiation therapy in treating patients with non-small cell lung cancer, small cell lung cancer, or neuroendocrine tumors that have spread from the original (primary) tumor to the brain (brain metastases). Berzosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving berzosertib together with radiation therapy may work better compared to standard of care treatment, including brain surgery and radiation therapy, in treating patients with non-small cell lung cancer, small cell lung cancer, or neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To conduct a phase 1 dose escalation trial in patients with brain metastases from non-small cell lung cancer (NSCLC) to determine the recommended phase 2 dose (RP2D) of twice weekly intravenous (i.v.) M6620 (VX-970, berzosertib) administered concurrent with conventionally fractionated whole brain radiotherapy (WBRT), with M6620 (VX-970, berzosertib) starting 18-30 hours after the first dose of radiation (but prior to the second fraction of radiation).

SECONDARY OBJECTIVES:

I. To estimate the incidence of >= grade 3 delayed neurological toxicity at 2, 4 and 6-months post-completion of whole-brain radiotherapy (for patients without intracranial progression).

II. To observe and record anti-tumor activity. IIa. To estimate the radiological response rates (RR) at 6 months including bi-directional and volumetric measurements of lesion size.

IIb. To estimate the intracranial 6-month progression-free survival (PFS).

EXPLORATORY/HYPOTHESIS GENERATING OBJECTIVES:

I. Changes in dynamic susceptibility contrast enhancement (DSC-magnetic resonance imaging [MRI]) perfusion and mean apparent diffusion coefficient (ADC) measurements in diffusion-weighted magnetic resonance imaging (DWI). (Group I) II. To measure cerebrospinal fluid (CSF) M6620 (VX-970, berzosertib) levels, tumor M6620 (VX-970, berzosertib) levels, and pATR T1989, pCHK1 S345 and RAD51 multiplex foci. (Group II) III. Changes in DSC-MRI perfusion and mean ADC measurements in DWI. (Group II)

OUTLINE: This is a dose-escalation study of berzosertib. Patients are assigned to 1 of 2 treatment groups.

GROUP I: Patients undergo whole-brain radiation therapy once daily (QD), 5 days a week for 15 fractions. Patients also receive berzosertib intravenously (IV) over 60-90 minutes twice a week, 18-30 hours after first radiation therapy. Treatment continues for 3 weeks in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive berzosertib IV over 60-90 minutes 2-4 hours prior to surgery. After surgery, patients undergo whole-brain radiation therapy and receive berzosertib as in Group I.

After completion of study treatment, patients are followed up every 2 months for 6 months, every 3-4 months for 6 months, then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed diagnosis of non-small cell lung cancer (NSCLC), including neuroendocrine tumors or small cell lung cancer (SCLC) who are being evaluated for palliative WBRT (with or without neurosurgical resection or stereotactic radiosurgery [SRS]) for radiologically or histologically diagnosed brain metastases presumed to be from the lung cancer are eligible for this Phase I study. Group 2 will only include NSCLC patients.
* Life expectance of greater than two months to allow completion of study treatment and assessment of dose-limiting toxicity
* Group 2 patients should have archived or fresh tumor tissue available from the non-craniotomy site and will have fresh tumor tissue available from the planned craniotomy
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of M6620 (VX-970, berzosertib) in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)

  * Note: though patients with ECOG performance status of 3 due to neurological deficits who are otherwise fit to receive systemic therapy per clinician assessments will be allowed
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* If no known liver metastases: total bilirubin < 1.5 x institutional upper limit of normal (ULN); if known liver metastases, then: total bilirubin < 2.5 x ULN
* If no known liver metastases: aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) < 2 x ULN; if known liver metastases, then: AST/SGOT of ALT/SGPT < 5 x ULN
* Creatinine within normal institutional limits for age OR creatinine clearance >= 45 mL/min/1.73 m^2 for patients with creatinine levels above ULN
* Negative serum or urine pregnancy test result for females of child bearing potential

  * The effects of M6620 (VX-970, berzosertib) on the developing human fetus are unknown. For this reason and because radiation therapy is known to have teratogenic potential, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of M6620 (VX-970, berzosertib) administration.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with 1-3 brain metastases, each < 3 cm by contrast MRI, with stable systemic disease and ECOG score of 0-2, who would otherwise be eligible for SRS/stereotactic radiation therapy (SRT) alone should not be enrolled into this study unless WBRT is recommended due to any medical reasons or logistic limitations as determined by the treating physician. Patients who develop recurrence post-SRS/SRT or surgery alone and are recommended WBRT will be eligible for the protocol.
* Greater than 1 cm mid-line shift, severe uncal herniation or significant hemorrhage/hydrocephalus (intra-lesional hemorrhage is acceptable). Patients with seizure at presentation who have been started on levetiracetam and have been stable for 48 hours prior to study registration are eligible at the discretion of treating physician
* Patients who have received systemic cytotoxic chemotherapy and/or, immunotherapy or other intravenous standard therapy for 2 weeks before initiation of planned WBRT, for oral targeted agents 3-7 days per clinician discretion or patients who have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or less from serious (CTCAE grade 3 or more) adverse events form the previously received agents. For any other investigational agents, at least 4 half-lives of the agent (6 weeks for nitrosoureas or mitomycin C) should have elapsed prior to starting study treatment
* Patients must not have received prior WBRT (previous SRS/SRT done at least 2 weeks from the planned start of WBRT is acceptable). Patients planned upfront to undergo SRS/SRT/fractionated boosts or neurosurgery after WBRT are not eligible; however, these treatments/procedures can be performed once the dose limiting toxicity (DLT) assessment has been completed, if felt clinically necessary
* Pregnant women are excluded from this study because M6620 (VX-970, berzosertib) as a deoxyribonucleic acid (DNA)-damage response (DDR) inhibitor may have the potential for teratogenic or abortifacient effects. Further, radiation therapy is known to have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with M6620 (VX-970, berzosertib), breastfeeding should be discontinued if the mother is treated with M6620 (VX-970, berzosertib).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to M6620 (VX-970, berzosertib).
* M6620 (VX-970, berzosertib) is primarily metabolized by cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); therefore, concomitant administration with strong inhibitors or inducers of CYP3A4 should be avoided. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference for a list of drugs to avoid or minimize use of. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product. Ongoing phenytoin should be either discontinued if clinically safe or transitioned to non-enzyme-inducing antiepileptics like levetiracetam with a 8-day washout period (half-life 18-22 hours, time to steady-state 4-8 days) prior to first dose of M6620 (VX-970, berzosertib) (7-days prior to WBRT).
* Patients needing more than 8 mg dexamethasone per day at the time of start of WBRT will not be eligible to participate in the study. However, patients will be allowed entry into the study if it is medically safe to reduce the daily dose of dexamethasone to 8 mg or less from the day of the start of WBRT. The dexamethasone dose for such patients may be increased beyond 8 mg per day during the course of treatment if medically necessary. This increased need for dose should be communicated to the study's principal investigator, Dr Mohindra at the University of Maryland.
* Uncontrolled intercurrent illness that would increase the risk of toxicity or limit compliance with study requirements. This includes but is not limited to, ongoing uncontrolled serious infection requiring i.v. antibiotics at the time of registration, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with M6620 (VX-970, berzosertib) and the uncertainties of any impact thereof on the radiation toxicities. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with known diagnoses that are associated with germline DDR defects such as Li Fraumeni syndrome and ataxia telangiectasia are excluded from the study as M6620 (VX-970, berzosertib) is a DDR inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2026-09-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pranshu Mohindra, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (9):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Case Western Reserve University, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - Dose Level 1: Patients undergo whole-brain radiation therapy Monday through Friday for 3 weeks for a total of 15 fractions. Patients also receive berzosertib 50 mg by infusion over 60-90 minutes twice a week, 18-30 hours after first radiation therapy.
- Group 1 - Dose Level 2: Patients undergo whole-brain radiation therapy Monday through Friday for 3 weeks for a total of 15 fractions. Patients also receive berzosertib 100 mg by infusion over 60-90 minutes twice a week, 18-30 hours after first radiation therapy.
- Group 2: Patients receive berzosertib at the identified dose in Group 1 by infusion over 60-90 minutes 2-4 hours prior to surgery. After surgery, patients undergo whole-brain radiation therapy Monday through Friday for 3 weeks for a total of 15 fractions. Patients also receive berzosertib at the dose identified in Group 1 by infusion over 60-90 minutes twice a week, 18-30 hours after first radiation therapy.
Period: Overall Study
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Started | 11 | 4 | 0
Completed | 9 | 2 | 0
Not Completed | 2 | 2 | 0
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Did not start treatment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was closed before enrolling to Group 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2 | Total
Number analyzed (Participants) | 11 | 4 | 0 | 15
Age, Continuous [Median (Full Range); unit: years] | 59 [51 to 78] | 63 [47 to 74] |  | 59 [47 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 |  | 9
  Male | 3 | 3 |  | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 11 | 4 |  | 15
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 1 | 1 |  | 2
  White | 10 | 3 |  | 13
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 4 |  | 15
Height [Median (Full Range); unit: centimeter (cm)] | 162.5 [150 to 187.9] | 179.2 [173 to 183] |  | 170 [150 to 187.9]
Weight [Median (Full Range); unit: kilogram (kg)] | 74.5 [59.4 to 105.7] | 69.3 [52.3 to 90.4] |  | 72.7 [52.3 to 105.7]
Body Surface Area [Median (Full Range); unit: meters squared (m^2)] | 1.9 [1.6 to 2.3] | 1.9 [1.6 to 2.1] |  | 1.9 [1.6 to 2.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-limiting Toxicity
Description: Defined as any grade 3 or more non-hematological toxicity requiring more than 5 day interruption in therapy or any grade 4 or higher hematological toxicity that is attributable to the berzosertib (M6620 [VX-970]) and/or whole brain radiotherapy
Time Frame: Up to 3 weeks after completing whole brain radiotherapy (WBRT)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2
Number analyzed (Participants) | 9 | 2
Participants
  Experiencing a dose limiting toxicity | 2 | 0
  Not experiencing a dose limiting toxicity | 7 | 2

2. Secondary Outcome: Incidence of Delayed Neurological Toxicity
Description: Assessed using Hopkins Verbal Learning Test-Revised. Incidence of events will be expressed as proportions with exact 95% confidence limits.
Time Frame: Up to 6-months post-completion of WBRT
Population: Not collected
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Changes in Quality of Life
Description: Measured by the Functional Assessment of Cancer Therapy-Brain. Descriptive statistics of the actual change scores will also be provided. The median change score and quartiles will be reported. Where relevant the proportion of patients experiencing a clinically significant change in score will be reported with 95% confidence limits.
Time Frame: Baseline to up to 6 months post-completion of WBRT
Population: Not collected
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Radiological Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR) is the disappearance of all target lesions; Partial Response (PR) is >=30% decrease in the sum of the target lesions; Disease Progression (PD) is >= 20% increase in the smallest sum of the target lesions; Stable Disease (SD) is between PR and PD.
Time Frame: 6 months
Population: Study was closed before enrolling to Group 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Number analyzed (Participants) | 9 | 2 | 0
Participants
  Complete response | 0 | 0 |
  Partial response | 0 | 0 |
  Stable disease | 3 | 0 |
  Disease progression or Death | 6 | 1 |
  No assessment | 0 | 1 |

5. Secondary Outcome: Intracranial Progression-free Survival (icPFS)
Description: Kaplan-Meier estimates of median icPFS will be calculated. Patients alive without intracranial progression at last follow-up will be censored at the date of the last radiologic assessment.
Time Frame: 6 months
Population: Not collected.
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Overall Survival (OS)
Description: Kaplan-Meier estimates of OS will be calculated. For calculation of OS, patients alive at last follow-up will be censored. Exploratory Cox regression analysis with M6620 (VX-970) dose as a covariate will be performed.
Time Frame: 12 months
Population: Study was closed before enrolling to Group 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Number analyzed (Participants) | 8 | 2 | 0
Participants
  Alive | 2 | 0 |
  Deceased | 6 | 0 |
  Not evaluable | 0 | 2 |

7. Other Pre Specified Outcome: Changes in Dynamic Susceptibility Contrast-magnetic Resonance Imaging Perfusion (Group I and II)
Description: Descriptive statistics of the actual change scores will also be provided. The median change score and quartiles will be reported. Where relevant the proportion of patients experiencing a clinically significant change in score will be reported with 95% confidence limits.
Time Frame: Baseline to up to 12 months
Population: Not collected
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Number analyzed (Participants) | 0 | 0 | 0

8. Other Pre Specified Outcome: Pharmacokinetic Characteristics of M6620 (VX-970) (Group II)
Description: Pharmacokinetics of the presence of M6620 (VX-970) in blood, CSF, and tissue will be assessed.
Time Frame: During surgery, pre-dose, and 2 hours and 50 minutes after start of M6620 (VX-970) infusion
Population: Not collected.
Arm/Group | Group 2
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Pharmacodynamic Properties of pATR T1989, pCHK1 S345 and RAD51 in Cerebrospinal Fluid (CSF) Post-M6620 (VX-970) Administration (Group II)
Time Frame: At 3 weeks post completion of WBRT
Population: Not collected
Arm/Group | Group 2
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Mean Apparent Diffusion Coefficient in Diffusion-weighted Magnetic Resonance Imaging (Group I and II)
Description: Descriptive statistics of the actual change scores will be provided.
Time Frame: Up to 12 months
Population: Not collected
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2 | Group 2
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Group 1 - Dose Level 1 | Group 1 - Dose Level 2
All-Cause Mortality (participants affected / at risk) | 7/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 5/9 | 0/2
Other Adverse Events (participants affected / at risk) | 9/9 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Dose Level 1 (N=9) | Group 1 - Dose Level 2 (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | NA
Anorexia (Metabolism and nutrition disorders) | 1 (1) | NA
Confusion (Psychiatric disorders) | 1 (1) | NA
Dehydration (Metabolism and nutrition disorders) | 1 (1) | NA
Otitis externa (Infections and infestations) | 1 (1) | NA
Platelet count decreased (Investigations) | 1 (1) | NA
Sepsis (Infections and infestations) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Dose Level 1 (N=9) | Group 1 - Dose Level 2 (N=2)
Agitation (Psychiatric disorders) | 1 (1) | 0
Alkaline phosphatase increased (Investigations) | 1 (3) | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0
Anemia (Blood and lymphatic system disorders) | 2 (6) | 0
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 0
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (2) | 0
Dizziness (Nervous system disorders) | 2 (2) | 0
Dysgeusia (Nervous system disorders) | 1 (1) | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0
Fatigue (General disorders) | 6 (8) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0
Mucosal infection (Infections and infestations) | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 5 (6) | 0
Paresthesia (Nervous system disorders) | 1 (1) | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 2 (4) | 0
Watering eyes (Eye disorders) | 1 (1) | 0
White blood cell count decreased (Investigations) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT02589522/Prot_SAP_000.pdf